CLINICAL TRIAL: NCT06121297
Title: A Phase 1/2, Open-label Study to Evaluate the Safety and Efficacy of Autologous CD19-specific Chimeric Antigen Receptor T Cells (CABA-201) in Subjects With Active Systemic Lupus Erythematosus
Brief Title: RESET-SLE: A Phase 1/2 Open-Label Study to Evaluate the Safety and Efficacy of CABA-201 in Subjects With Active Systemic Lupus Erythematosus
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Cabaletta Bio (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CAB-201-001
Record Dates: First submitted 2023-10-23; First posted 2023-11-07 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Systemic Lupus Erythematosus; Lupus Nephritis
Keywords: CABA-201; Autoimmune Disease; Anti-CD19 CAR-T therapy; Cellular Therapy; Systemic Lupus Erythematosus; Lupus Nephritis
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Lupus Nephritis; Autoimmune Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CABA-201 with FLU/CY Preconditioning (Experimental): LN Cohort: Infusion of CABA-201 with preconditioning in subjects with LN
  Non-renal SLE Cohort: Infusion of CABA-201 with preconditioning in subjects with non-renal SLE who do not meet criteria for inclusion in the LN cohort
  Expansion Cohort: Infusion of CABA-201 with preconditioning in subjects with LN and SLE
  Interventions: Biological: CABA-201
- CABA-201, No Preconditioning (Experimental): Infusion of CABA-201 with no preconditioning in subjects with LN and non-renal SLE
  Interventions: Biological: CABA-201

INTERVENTIONS:
Biological: CABA-201 — Single intravenous infusion of CABA-201 at a single dose level following preconditioning with fludarabine and cyclophosphamide
  Arms: CABA-201 with FLU/CY Preconditioning
Biological: CABA-201 — Single intravenous infusion of CABA-201 at escalating dose levels without preconditioning
  Arms: CABA-201, No Preconditioning

SUMMARY:
RESET-SLE: A Phase 1/2 Open-Label Study to Evaluate the Safety and Efficacy of CABA-201 in Subjects With Active Systemic Lupus Erythematosus

DETAILED DESCRIPTION:
Systemic lupus erythematosus (SLE) is a chronic autoimmune disorder characterized by autoantibody production and abnormal B cell function. SLE presents with fluctuating severity and may cause tissue damage in a variety of organs over time. Lupus nephritis (LN) (renal involvement) is a common severe manifestation of SLE, which can lead to significant morbidity and mortality. This study is being conducted to evaluate the safety and efficacy of an investigational cell therapy, CABA-201, also called resecabtagene autoleucel, or "rese-cel". Rese-cel can be given to patients with either LN or SLE without renal involvement, in two separate parallel cohorts, who have active disease. Initially a single dose of CABA-201 in patients pretreated with a standard regimen including cyclophosphamide (CY) and fludarabine (FLU), will be evaluated. In addition, escalating doses of CABA-201 will be evaluated in patients without CY and FLU pretreatment.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 and ≤65
* A clinical diagnosis of SLE, based on the 2019 European League Against Rheumatism (EULAR)/American College of Rheumatology (ACR) classification criteria for adult SLE.
* Positive antinuclear antibody (ANA) titer or anti-dsDNA antibody at screening.
* For LN subjects only, active, biopsy-proven LN class III or IV, with or without the presence of class V, according to 2018 Revised International Society of Nephrology/Renal Pathology Society (ISN/RPS) criteria
* For non-renal SLE subjects only: Active, moderate to severe SLE

Exclusion Criteria:

* Contraindication to leukapheresis
* History of anaphylactic or severe systemic reaction to fludarabine, cyclophosphamide or any of their metabolites
* Active infection requiring medical intervention at screening
* Current symptoms of severe, progressive, or uncontrolled renal, hepatic, hematological, gastrointestinal, pulmonary, psychiatric, cardiac, neurological, or cerebral disease, including severe and uncontrolled infections, such as sepsis and opportunistic infections.
* Concomitant medical conditions that, in the opinion of the investigator, might place the subject at unacceptable risk for participation in this study, interfere with the assessment of the effects or safety of the investigational product or with the study procedures
* For LN subjects only: The presence of kidney disease other than active lupus nephritis
* Previous CAR T cell therapy
* Prior solid organ (heart, liver, kidney, lung) transplant or hematopoietic cell transplant.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2024-02-16 (Actual); Primary Completion 2029-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
To evaluate incidence of adverse events | Up to 28 days after CABA-201 infusion

SECONDARY OUTCOMES:
To evaluate adverse events and laboratory abnormalities | Up to 156 weeks
  Incidence and severity of AEs, including changes in laboratory values and vital signs
To characterize the pharmacodynamics (PD) | Up to 156 weeks
  Levels of B cells in the blood
To characterize the pharmacokinetics (PK) | Up to 156 weeks
  Levels of CABA-201-positive T cells in the blood
To evaluate disease related biomarkers | Up to 156 weeks
  Levels of C3, C4, and CH50 in serum
To evaluate disease related biomarkers | Up to 156 Weeks
  Levels of anti-double stranded DNA (anti-dsDNA) in serum
To evaluate efficacy | Up to 156 Weeks
  Complete renal response rates (in subjects with LN)
To evaluate efficacy | Up to 156 weeks
  SRI-4, BICLA and DORIS remission and LLDAS response rates

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Chair — Cabaletta Bio
Locations (23):
- United States (21):
  - University of California Irvine, Orange, California
  - UC Davis Health, Sacramento, California
  - Yale University, New Haven, Connecticut
  - University of Florida Health, Gainesville, Florida
  - Mayo Clinic, Jacksonville, Florida
  - Emory University, Atlanta, Georgia
  - Northwestern Memorial Hospital, Chicago, Illinois
  - The University of Chicago Medical Center, Chicago, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - Tufts Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Boston Children's Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - UMass Memorial Hospital, Worcester, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - Columbia University Irving Medical Center, New York, New York
  - University of Rochester, Rochester, New York
  - UNC Chapel Hill, Chapel Hill, North Carolina
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Texas MD Anderson Cancer Center, Houston, Texas
- Maisonneuve-Rosemont Hospital, Montreal, Quebec, Canada
- Clinica Universitaria de Navarra, Pamplona, Navarre, Spain

IPD SHARING:
Plan to Share IPD: No